CLINICAL TRIAL: NCT03781583
Title: Smart Head Mounted Display (smartHMD) for Improved Mobility
Brief Title: SmartHMD for Improved Mobility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: James Weiland (Other)
Responsible Party: Sponsor-Investigator, James Weiland, Professor of Biomedical Engineering, University of Michigan
Organization: University of Michigan (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HUM00141598
Record Dates: First submitted 2018-12-12; First posted 2018-12-20 (Actual); Results first posted 2024-12-12 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Low Vision; Orientation; Mobility Limitation; Navigation, Spatial; Visual Impairment
MeSH Terms: conditions — Vision, Low; Orientation, Spatial; Mobility Limitation; Spatial Navigation; Vision Disorders

STUDY DESIGN:
Intervention Model Description: Testing will be done in three conditions: baseline (no HMD), sham (smartHMD worn but not active), and smartHMD (smartHMD worn and active)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (4):
- Outdoor and ODG (Experimental): Participants used the first version of the SmartHMD device, which used custom software running on commercially available ODG R7 smart glasses and accompanying earbuds. Participants used the device to navigate across an outdoor crosswalk.
  Interventions: Device: SmartHMD version 1
- Indoor and Laptop (Experimental): Participants use the second version of the SmartHMD device, which uses RGB-D smart glasses, custom software running on a laptop, and bone-conducting earphones. Participants use the device to locate the door within an indoor course.
  Interventions: Device: SmartHMD version 2
- RGBD & Jetson - Indoor Course (Experimental): Participants use a new iteration of the SmartHMD device, which uses RGB-D smart glasses, bone-conducting earphones, a Jetson mobile computer, and custom software. Participants use the device to navigate their way through an indoor course.
  Interventions: Device: SmartHMD version 3
- RGBD & Jetson - Outdoor Crosswalk (Experimental): Participants use the SmartHMD device, which uses RGB-D smart glasses, bone-conducting earphones, a Jetson mobile computer, and a specific version of custom software. Participants use the device to navigate their way through an outdoor crosswalk.
  Interventions: Device: SmartHMD version 4

INTERVENTIONS:
Device: SmartHMD version 1 — First version of the SmartHMD device, which used custom software running on commercially available ODG R7 smart glasses and accompanying earbuds.
  Arms: Outdoor and ODG
Device: SmartHMD version 2 — Second version of the SmartHMD device, which uses RGB-D smart glasses, custom software running on a laptop, and bone-conducting earphones.
  Arms: Indoor and Laptop
Device: SmartHMD version 3 — Third iteration of the SmartHMD device, which uses RGB-D smart glasses, bone-conducting earphones, a Jetson mobile computer, and custom software.
  Arms: RGBD & Jetson - Indoor Course
Device: SmartHMD version 4 — Fourth iteration of the SmartHMD device, which uses RGB-D smart glasses, bone-conducting earphones, a Jetson mobile computer, and a specific version of custom software.
  Arms: RGBD & Jetson - Outdoor Crosswalk

SUMMARY:
The National Eye Institute estimated about 3 million people over age 40 in the US had low vision in 2010 and projects an increase to nearly 5 million in 2030 and 9 million in 2050. Current assistive technologies are a patchwork of mostly low-technology aids with limited capabilities that are often difficult to use, and are not widely adopted. This shortfall in capabilities of assistive technology often stems from lack of a user-centered design approach and is a critical barrier to improve the everyday activities of life (EDAL) and the quality of life (QOL) for individuals with low vision.

An intuitive head mounted display (HMD) system on enhancing orientation and mobility (O&M) and crosswalk navigation, could improve independence, potentially decrease falls, and improve EDAL and QOL. The central hypothesis is that an electronic navigation system incorporating computer vision will enhance O&M for individuals with low vision. The goal is to develop and validate a smartHMD by incorporating advanced computer vision algorithms and flexible user interfaces that can be precisely tailored to an individual's O&M need. This project will address the specific question of mobility while the subject crosses a street at a signaled crosswalk. This is a dangerous and difficult task for visually impaired patients and a significant barrier to independent mobility.

DETAILED DESCRIPTION:
This study was originally intended as a single-arm study. Early results and unanticipated events related to component availability made it clear that multiple configurations of the device would be necessary to produce a functional device. Therefore, the study was split into multiple cohorts representing each iteration of the device and testing process, as follows:

As the trial progressed, the participants recruited were consistently unable to perform tasks without smartHMD. This is due to the recruitment of participants with severe vision loss. Due to this finding, data was only acquired when participants used the smartHMD when active instead of collecting data with and without the system being active.

The participants performed a subset of experiments due to time constraints. Some performed only outdoor trials; some performed only indoor trials; others performed both. The outcome measures depend on which experiments were performed.

After the first test involving the initial three participants, the ODG system became unsupported by the company that produced the device. In response, the study team developed a prototype system (RGBD), which was used in the ODG system's place for the remaining tests. The RGBD was initially used indoors with laptop and subsequently outdoors with mobile hardware and new software.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with low vision
* Self reported difficulty with mobility and finding doors (either indoors or outdoors) and using signalized crosswalks.
* Ability to cooperate for tests
* Able to participate in all visits

Exclusion Criteria:

* Unable to use head mounted display technology
* Unstable age-related macular degeneration within the past 3 months
* Unstable diabetic retinopathy within the past 3 months
* Unstable diabetes within the past 3 months
* Ocular infection or ocular inflammation in the past 3 months
* Ocular trauma within the past 6 months
* Intraocular surgery within 6 months
* Optical coherence tomography retinal findings of concern to investigator for unstable vision during the study
* Women who are pregnant (due to risk of falls and change in gait).
* Uncontrolled seizure disorder in the past 6 months
* Cerebrovascular accident occurring in the past 6 months
* Parkinson disease or neurological condition that limits mobility
* Alzheimer disease or other forms of dementia
* Conditions of concern to investigator that would confound orientation and mobility, such as severe arthritis, pain that limits ambulatory activities, or orthopedic surgery (e.g., hand, arm, shoulder, knee, or hip surgery within 12 months)

Ages: 14 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-04-26 (Actual); Primary Completion 2022-11-07 (Actual); Study Completion 2022-11-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Weiland, PhD, Principal Investigator — University of Michigan
Locations (1):
- North Campus Research Complex, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 21 people consented, 2 individuals failed post start-up screening, and 1 never came in for any assignment. That brings the 21 consented to 18.
  Participants could consent and enroll in multiple cohorts, reconsenting for each cohort in which they participated. The numbers shown in each arm represent each individual who initially enrolled in that cohort. Some continued on to participate in further tests, but no participant appears in more than one arm in Participant Flow.
Groups:
- Cohort A: Outdoor and ODG: This cohort began their participation by testing this iteration of the SmartHMD device. Some participants, as shown below via milestones, also participated in subsequent tests.
  SmartHMD version 1 assessed with Outdoor Crosswalk Test: Participants used the first version of the SmartHMD device, which used custom software running on commercially available ODG R7 smart glasses and accompanying earbuds. Participants used the device to navigate across an outdoor crosswalk.
- Cohort B: Indoor and Laptop: This cohort began their participation by testing this iteration of the SmartHMD device. Some participants, as shown below via milestones, also participated in subsequent tests.
  SmartHMD version 2 assessed with Indoor Door Location Test: Participants use the second version of the SmartHMD device, which uses RGB-D smart glasses, custom software running on a laptop, and bone-conducting earphones. Participants use the device to locate the door within an indoor course.
- Cohort C: RGBD & Jetson - Indoor Course: This cohort began their participation by testing this iteration of the SmartHMD device. Some participants, as shown below via milestones, also participated in subsequent tests.
  SmartHMD assessed with Indoor Course: Participants use a new iteration of the SmartHMD device, which uses RGB-D smart glasses, bone-conducting earphones, a Jetson mobile computer, and custom software. Participants use the device to navigate their way through an indoor course.
- Cohort D: RGBD & Jetson - Outdoor Crosswalk: This cohort began their participation by testing this iteration of the SmartHMD device.
  SmartHMD assessed with outdoor crosswalk: Participants use the SmartHMD device, which uses RGB-D smart glasses, bone-conducting earphones, a Jetson mobile computer, and a specific version of custom software. Participants use the device to navigate their way through an outdoor crosswalk.
Period: Overall Study
Arm/Group | Cohort A: Outdoor and ODG | Cohort B: Indoor and Laptop | Cohort C: RGBD & Jetson - Indoor Course | Cohort D: RGBD & Jetson - Outdoor Crosswalk
Started (started means first participation was with this intervention and for this form of test) | 4 | 5 | 8 | 1
Participated and Completed Indoor Doorfinding Test | 1 | 3 | 0 | 0
RGBD & Jetson Test | 0 | 2 | 8 | 0
RGBD Outdoor Crosswalk Test | 0 | 1 | 1 | 1
Completed (This row shows those who began in that arm and completed its test, but for any specific test other than the first (pre-pandemic crosswalk), the number of people who completed that test can be read by adding across the row of the milestone.) | 2 | 3 | 8 | 1
Not Completed | 2 | 2 | 0 | 0
Not completed — Technical issue prevents the device from starting properly | 1 | 0 | 0 | 0
Not completed — Technology did not work for that person in that environment | 1 | 0 | 0 | 0
Not completed — Participant was not sufficiently visually impaired | 0 | 1 | 0 | 0
Not completed — Pilot test of course took place in different location, data not comparable to other participant data | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The numbers shown in each arm below represent one person beginning in that cohort.
Groups:
- Cohort C: RBDG & Jetson -Indoor: This cohort began their participation by testing this iteration of the SmartHMD device. Some participants, as shown below via milestones, also participated in subsequent tests.
  SmartHMD assessed with Indoor Course: Participants use a new iteration of the SmartHMD device, which uses RGB-D smart glasses, bone-conducting earphones, a Jetson mobile computer, and custom software. Participants use the device to navigate their way through an indoor course.
- Total: Total of all reporting groups
Arm/Group | Cohort A: Outdoor and ODG | Cohort B: Indoor and Laptop | Cohort C: RBDG & Jetson -Indoor | Cohort D: RGBD & Jetson - Outdoor Crosswalk | Total
Number analyzed (Participants) | 4 | 5 | 8 | 1 | 18
Age, Customized [Count of Participants; unit: Participants] — Population: Age information was not collected
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 5 | 4 | 1 | 10
  Male | 4 | 0 | 4 | 0 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 4 | 5 | 8 | 1 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 4 | 5 | 8 | 1 | 18
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 | 5 | 8 | 1 | 18
Preferred Walking Speed [Mean (Full Range); unit: meters/second] — Baseline Measure data was only collected for tests C and D. Population: Baseline Measure data was only collected for tests C and D.
  meters/second
    Preferred walking speed of those testing the indoor course (Test C): number analyzed (Participants) | 0 | 2 | 8 | 0 | 10
    Preferred walking speed of those testing the indoor course (Test C) |  | .622 [.427 to .817] | .968 [.76 to 1.156] |  | .899 [.427 to 1.156]
    Preferred walking speed of those testing the outdoor course (Test D): number analyzed (Participants) | 0 | 1 | 1 | 1 | 3
    Preferred walking speed of those testing the outdoor course (Test D) |  | .817 [.817 to .817] | 0.76 [.76 to 0.76] | 1.15 [1.15 to 1.15] | .909 [.76 to 1.15]

OUTCOME MEASURES:

1. Primary Outcome: Time-to-Complete
Description: Duration from start of trial to subject completing their assigned task (seconds).
Time Frame: 2 hours
Population: Data are not included for those participants who did not show up, equipment malfunctions or persons unable to complete the task.
Measure: Mean (Full Range); unit: Seconds
Groups:
- Study Participants: Participants in this study could participate in multiple tests within the study. The total number in this arm reflects the number of unique participants. The number analyzed within each test reflects the number of participants who participated in that specific test and for whom usable data was collected. Some participants did participate in more than one test.
Arm/Group | Study Participants
Number analyzed (Participants) | 16
Seconds
  Outdoor Crosswalk with ODG Test: number analyzed (Participants) | 2
  Outdoor Crosswalk with ODG Test | 14.75 [13 to 17]
  Indoor Door Finding Test: number analyzed (Participants) | 4
  Indoor Door Finding Test | 32.75 [18 to 55]
  Indoor Course Navigation Test: number analyzed (Participants) | 10
  Indoor Course Navigation Test | 148.17 [40 to 479]
  Outdoor Crosswalk with RGBD, Jetson New Software Test: number analyzed (Participants) | 3
  Outdoor Crosswalk with RGBD, Jetson New Software Test | 17.3 [12.15 to 20.2]

2. Secondary Outcome: Percentage of Preferred Walking Speed
Description: Percentage of preferred walking speed is a measure of how fast the participant is walking relative to their natural (or preferred) walking speed. Measure preferred walking speed was measured by having them walk with a researcher in an open area. Percentage preferred walking speed was obtained by dividing the measured walking speed during a trial by the preferred walking speed.
Time Frame: 2 hours
Population: Participants in this study could participate in multiple tests within the study. The total number in this arm reflects the number of unique participants. The number analyzed within each test reflects the number of participants who participated in that specific test and for whom usable data was collected. Some participants did participate in more than one test.
Measure: Mean (Full Range); unit: percentage of preferred walking speed
Arm/Group | Study Participants
Number analyzed (Participants) | 11
percentage of preferred walking speed
  RGBD & Jetson indoor test: number analyzed (Participants) | 10
  RGBD & Jetson indoor test | 67.2 [26.6 to 150]
  RGBD and Jetson Outdoor Crosswalk test: number analyzed (Participants) | 3
  RGBD and Jetson Outdoor Crosswalk test | 95.76 [86.5 to 104.25]

3. Secondary Outcome: Number of Unintended Contacts With Obstacles and Walls
Description: This outcome measure only applies to the RGBD & Jetson Indoor Test, as there were no walls/obstacles relevant in the other tests.
Time Frame: 2 hours
Population: This includes all participants who completed this test and for whom usable data was collected.
Measure: Mean (Full Range); unit: Count of contacts
Groups:
- RGBD & Jetson Test (Indoor Course): Course: Participants use a new iteration of the SmartHMD device, which uses RGB-D smart glasses, bone-conducting earphones, a Jetson mobile computer, and custom software. Participants use the device to navigate their way through an indoor course.
Arm/Group | RGBD & Jetson Test (Indoor Course)
Number analyzed (Participants) | 10
Count of contacts | 0 [0 to 0]

4. Secondary Outcome: Number of Incorrect Turns
Description: Number of incorrect turns or responses to device cues during testing.
Time Frame: 2 hours
Population: Data was only collected for the RGBD & Jetson indoor test and the RGBD and Jetson Outdoor Crosswalk test
Measure: Median (Full Range); unit: Count of incorrect turns
Arm/Group | Study Participants
Number analyzed (Participants) | 11
Count of incorrect turns
  RGBD & Jetson indoor test: number analyzed (Participants) | 10
  RGBD & Jetson indoor test | 0 [0 to 7]
  RGBD and Jetson Outdoor Crosswalk test: number analyzed (Participants) | 3
  RGBD and Jetson Outdoor Crosswalk test | 1 [0 to 8]

5. Secondary Outcome: Number of Interventions
Description: Upon real-world application of the study protocol, the outcome measure originally conceived of as "requests for assistance" became pragmatically inseparable from "number of interventions" by study staff. Therefore, the two measures have been combined and are presented here as "number of interventions". The types of assistance requested could not be categorized, as they were not collected.
Time Frame: 2 hours
Population: Data was only collected for the RGBD & Jetson indoor test and the RGBD and Jetson Outdoor Crosswalk test
Measure: Median (Full Range); unit: Counts of interventions
Arm/Group | Study Participants
Number analyzed (Participants) | 11
Counts of interventions
  Indoor Course Navigation Test: number analyzed (Participants) | 10
  Indoor Course Navigation Test | 0 [0 to 5]
  Outdoor Crosswalk with RGBD, Jetson New Software Test: number analyzed (Participants) | 3
  Outdoor Crosswalk with RGBD, Jetson New Software Test | 0 [0 to 3]

ADVERSE EVENTS:
Time Frame: AEs could have been collected during on-site participation, up to two hours. Follow-up calls took place two weeks later, during which participants could have reported AEs.
Groups:
- Outdoor and ODG Test Participants: SmartHMD version 1 assessed with Outdoor Crosswalk Test: Participants used the first version of the SmartHMD device, which used custom software running on commercially available ODG R7 smart glasses and accompanying earbuds. Participants used the device to navigate across an outdoor crosswalk.
- Cohort B: Indoor and Laptop Test Participants: SmartHMD version 2 assessed with Indoor Door Location Test: Participants use the second version of the SmartHMD device, which uses RGB-D smart glasses, custom software running on a laptop, and bone-conducting earphones. Participants use the device to locate the door within an indoor course.
- Cohort C: RGBD & Jetson - Indoor Test Participants: SmartHMD assessed with Indoor Course: Participants use a new iteration of the SmartHMD device, which uses RGB-D smart glasses, bone-conducting earphones, a Jetson mobile computer, and custom software. Participants use the device to navigate their way through an indoor course.
- Cohort D: RGBD & Jetson - Outdoor Crosswalk Test Participants: SmartHMD assessed with outdoor crosswalk: Participants use the SmartHMD device, which uses RGB-D smart glasses, bone-conducting earphones, a Jetson mobile computer, and a specific version of custom software. Participants use the device to navigate their way through an outdoor crosswalk.
  Participants use the device to navigate their way through an outdoor crosswalk.
Arm/Group | Outdoor and ODG Test Participants | Cohort B: Indoor and Laptop Test Participants | Cohort C: RGBD & Jetson - Indoor Test Participants | Cohort D: RGBD & Jetson - Outdoor Crosswalk Test Participants
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/6 | 0/10 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/6 | 0/10 | 0/3
Other Adverse Events (participants affected / at risk) | 0/4 | 0/6 | 0/10 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-29): https://cdn.clinicaltrials.gov/large-docs/83/NCT03781583/Prot_SAP_000.pdf